CLINICAL TRIAL: NCT06340074
Title: Helping Educational Leadership Mobilize Evidence (HELM): An Organizational Intervention to Promote Strategic Implementation in Schools
Brief Title: Helping Educational Leadership Mobilize Evidence
Acronym: HELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Aaron Lyon, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00010282
Record Dates: First submitted 2024-03-21; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Behavior, Child
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HELM (Experimental): Behavioral: HELM
  HELM is a 9-month, data-driven organizational and leadership implementation strategy.
  Interventions: Behavioral: HELM
- Implementation Attention Control (IAC) (Placebo Comparator): Behavioral: Implementation Attention Control (IAC)
  Schools assigned to the IAC condition received an online, self-paced, independent studies program broadly focused on leadership and management.
  Interventions: Behavioral: Implementation Attention Control (IAC)

INTERVENTIONS:
Behavioral: HELM — HELM is a 9-month, data-driven organizational and leadership implementation strategy that entails eight core components: 1) Assessment and Feedback. 2) Initial Training. 3) Leadership Development Plan. 4) Individual Coaching. 5) Group Coaching. 6) Organizational Strategy Development. 7) Professional Learning Collaboratives. 8) Graduation.
  Arms: HELM
Behavioral: Implementation Attention Control (IAC) — Schools assigned to the IAC condition received an online, self-paced, independent studies program broadly focused on leadership and management. The program did not specifically discuss implementation leadership or climate. The program included four content modules hosted on a web-based learning portal: 1) Motivating and Engaging Employees, 2) Authentic Leadership, 3) Managing Diverse Teams, and 4) Fostering an Idea Culture. Each module consisted of one content-specific 60-minute webinar.
  Arms: Implementation Attention Control (IAC)

SUMMARY:
Many universal, evidence-based prevention practices (EBPPs) have been developed to prevent SEB problems, typically in elementary schools, but progress toward widespread implementation has been slow and few efforts have been made to develop and test interventions to enhance EBPP implementation in schools. Schools leaders (e.g., principals) are key to decision making and implementation of EBPPs, and their leadership has been shown to be consistently linked to student outcomes through their intentional efforts to support teacher adoption and use of innovative programs. Helping Educational Leaders Mobilize (HELM) Evidence is a pragmatic, multifaceted, organizationally-focused implementation strategy targeting the implementation leadership and implementation climate of school buildings (through principals) to enhance the adoption and delivery of EBPPs in elementary schools. This pilot study, part of the larger HELM project to adapt and test the strategy based on an existing leadership intervention, Leadership and Organizational Change for Implementation (LOCI), will be implemented in the context of Positive Greetings at the Door (PGD), a universal school-based EBPP previously demonstrated to reduce disruptive behavior and increase academic engagement.

ELIGIBILITY:
Inclusion Criteria:

* Being a K-5th elementary school
* Being a K-5th principal or assistant principal at an elementary school
* Being a K-5th grade teacher, paraeducator, or specialist (e.g., reading) at an elementary school, and not a teacher in a special education-only classroom

Exclusion Criteria:

* School building or teacher that is currently implementing PGD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Proximal Outcome: Strategic Implementation Leadership | Baseline, 4-months, 8-months
  The School Implementation Leadership Scale (SILS) is an 25-item scale that assesses the degree to which a school's leader is perceived to engage in eight specific behaviors that are supportive of EBP implementation which both principals and educators complete. The eight subscales include: 1) supportive; 2) perseverant; 3) communication; 4) proactive; 5) availability; 6) knowledgeable; 7) vision/mission; and 8) distributed leadership.
Proximal Outcome: Strategic Implementation Climate | Baseline, 4-months, 8-months
  The School Implementation Climate Scale (SICS) is an 21-item scale for principals' and educators' shared perceptions of the policies, practices, and procedures that are expected, rewarded, and supported. The six subscales include: 1) focus on EBPs; 2) educational support for EBPs; 3) recognition for EBPs; 4) use of data to support EBPs; 5) existing supports to deliver EBPs; and 6) integration of EBPs.
Proximal Outcome: Implementation Citizenship Behavior | Baseline, 4-months, 8-months
  The School Implementation Citizenship Behavior Scale (SICBS) is a 12-item rating scale that measures principals' and educators' perceptions regarding how educators engage with EBPs within their specific school context. The four subscales include: 1) helping others; 2) keeping informed; 3) taking Initiative; and 4) advocacy.
Proximal Outcome: Implementation Initiative Stability | Baseline, 4-months, 8-months
  A modified version of the 8-item Commitment to Organizational Change Scale (COCS) will measure principals' and educators' perceptions of implementation initiative stability. Subscales include: Affective Commitment and Normative Commitment.
Implementation Outcome: Fidelity and Sustainment - Observed | 2-months, 2.5-months, 3-months, 3.5-months, 4-months, 4.5-months, 5-months, 6-months, 7-months, 8-months
  Assitant principals will be trained to conduct PGD fidelity observations and complete three PGD observations biweekly (October - December) and monthly (January - May) over the course of the school year. Minimum Score 0, Maximum Score 6. Higher Scores mean better outcome.
Implementation Outcome: Fidelity and Sustainment - Self Report | 4-months, 8-months
  A self-report fidelity rating scale will be used to capture adherence to delivering core PGD practices as planned. Educators will complete the rating scale at the mid-year and end-of-year assessments. Minimum Score 0, Maximum Score 4. Higher Scores mean better outcome.
Implementation Outcome: Reach | 9-months
  Reach will be computed using the fidelity data to determine the proportion of students who are receiving PGD practices. The number of general education teachers who are implementing PGD divided by the total number of teachers who have received PGD training.
Implementation Outcome: Facilitators and Barriers to Implementation | 9-months
  A qualitative interview for HELM participants will explore: (1) potential changes to HELM (e.g., "What parts of HELM could be improved to increase its appropriateness to schools?"); (2) opportunity costs of participating (e.g., "Were there any activities you wanted to do but could not because of participation in HELM?"); and (3) unintended consequences.
Implementation Outcome: Implementation Cost | 9-months
  Costs of (1) delivering the HELM intervention to augment PGD implementation, as well as (2) implementation as usual, will be calculated using standard average weighted cost metrics. Inputs will include time, supplies, travel, overhead, and costs associated with HELM training/coaching meetings, including pre-work, scheduling, and attending meetings.

SECONDARY OUTCOMES:
Student Educational Outcomes | 9-months
  Schools will complete a survey on student educational outcomes for the year, including questions related to grades (GPA) and standardized test scores. There is no reporting on a scale.
Student Behavioral Outcomes | 4-months, 8-months
  Modified Direct Behavior Rating Scale - A modified version of the Direct Behavior Rating Scale will be given to educators to assess their classroom's on-task behavior, prosocial behavior, ability to follow directions the first time, and disruptive behavior. These questions all are part of the same scale that ask the proportion of time their students spent doing each in the first five minute of class (0-100%) and proportion of time their students spent doing each the whole day (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School Mental Health Assessment, Research, and Training (SMART) Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained during the HELM study will be provided to researchers who have demonstrated an academic interest in educational services, in-school mental health services, or in implementation sciences. Outside investigators who wish to use the data set to answer new research questions may also submit data analysis concept proposals for consideration by the PI on a case-by-case basis. The PI will review the proposal and will provide those who submit scientifically rigorous and promising proposals access to the data repository to address their research questions. This will ensure that the data resources of the proposed study will provide the greatest possible benefit to the scientific community. Data samples that may be shared will be coded based on study design, and all personal health and identifying will be removed. Prerequisite to data sharing, the PI will require applicable agreements (i.e., data transfer agreements) with the requesting entity.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted to the PI starting 6 months after initial publication of the primary findings. The PI will continue to accept requests for those findings for 24 months following the end-date of the awarded grant.
Access Criteria: Access to study data can be requested by any qualified researchers who are engaging in independent scientific research, with approval dictated by the PI. Acceptance of data sharing will only be done following review of a sharing agreement.

REFERENCES:
- [Derived] Locke J, Corbin CM, Goosey R, Collins VK, Ehrhart MG, Hatch K, Espeland C, Lyon AR. Not getting better but not getting worse: A cluster randomized controlled pilot trial of a leadership implementation strategy. Implement Res Pract. 2025 Jan 29;6:26334895241312405. doi: 10.1177/26334895241312405. eCollection 2025 Jan-Dec. PMID 39881952